CLINICAL TRIAL: NCT06829121
Title: Ultrasound-based Morphometry for the Development of Diagnostic and Prognostic Markers in Current and Chronic Diseases
Status: Completed | Type: Observational
Sponsor: Universitatsmedizin Mainz - 1. Medizinische Klinik (Other)
Responsible Party: Principal Investigator, Wolfgang Maximilian Kremer, Senior physician, Universitatsmedizin Mainz - 1. Medizinische Klinik
Other Study IDs: 2020-15174
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound; Sarcopenia; Muscle Loss
Keywords: muscle measurement by ultrasound; evaluation of muscle mass
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ultrasound patients: Patients who receive a standard ultrasound also get a measurement of the musculature.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — The thickness of the psoas muscle and the musculus quadriceps femoris will be measured by ultrasound

SUMMARY:
Frailty or debility is a geriatric syndrome that primarily affects older patients, but also patients with severe illnesses. It is particularly common among oncology patients, but also among patients with gastrointestinal diseases such as liver cirrhosis or pancreatitis. Sarcopenia, a component of frailty, is defined as a loss of muscle quantity, quality and function. Currently, complex methods such as CT or bioimpedance measurement are available. However, simpler techniques such as ultrasound-based measurement could be alternatives, but require further validation.

The aim of this project is to be able to estimate the prognosis of patients at an early stage by measuring sarcopenia using sonography.

DETAILED DESCRIPTION:
Frailty is a well-known syndrome that has a negative impact on many diseases and the course of disease. Patients affected by frailty are particularly vulnerable due to their inadequate ability to deal with extrinsic and intrinsic stress factors. The prevalence of frailty increases with age, affecting 15% of people over the age of 65 and 25% of people over the age of 80.

Frailty is the end result of an interplay between malnutrition, cognitive impairment and muscle wasting. Each of these factors can be further examined and measured, but they also influence each other. In particular, reduced muscle mass and muscle function have been associated with poor quality of life and a worse course of disease. Sarcopenia is therefore becoming an increasingly important factor in various disease patterns and should be monitored further. Muscle wasting and sarcopenia have multifactorial causes. Physical inactivity, chronic inflammation associated with chronic diseases, and malnutrition are particularly noteworthy in this context. Cross-sectional measurement of several muscles at the level of the lumbar vertebrae (L3), normalized to body size, and dual-energy X-ray absorptiometry are currently the most commonly used techniques for measuring sarcopenia. However, the measurements require complex equipment and procedures. In addition, radiological imaging is costly and causes radiation exposure. Therefore, attempts have been made in the past to simplify the measurements. Sonographic measurement is a practical alternative. Many different muscle groups are accessible to ultrasound. In particular, the thigh muscles and the psoas major muscle can be easily visualized sonographically. The sonographic assessment of the psoas muscle area index (PMAI) and the thigh muscle thickness index (TMTI) are approaches for bedside morphometry that the investigators use primarily.

Sarcopenia needs to be further investigated and included in the evaluation of therapeutic concepts. Recently, Zhang et al. showed that radiologically measured reduced psoas muscle mass was associated with poorer overall survival in HCC patients. Furthermore, it has been suggested several times that sarcopenia should be integrated into the MELD classification for liver transplantation. The investigators were also recently able to show in a cohort of COVID-19 patients that reduced muscle mass was associated with a poorer disease course during the pandemic.

The investigators expect sonographic measurements of the musculature to provide a better assessment of prognosis, quality of life and functional results under therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive a planned ultrasound examination as part of their outpatient or inpatient evaluation during the planned period.
* All patients over 18 years of age.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients unable to give consent.
* Patients with neuromuscular disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients treated at the First Medical Clinic of the University Medical Center in Mainz who are scheduled to undergo a planned ultrasound examination.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Complication | From date of inclusion until the date of first documented decompensation or death from any cause, whichever came first, assessed up to two years
  Number of participants with decompensation of the underlying disease (e.g. liver cirrhosis: hydropic decompensation) or death

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Maximilian Kremer WMK Kremer, MD, Principal Investigator — Universitatsmedizin Mainz
Locations (1):
- Universitatsmedizin Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The data will be published as part of publications if necessary.

REFERENCES:
- [Background] Hari A, Berzigotti A, Stabuc B, Caglevic N. Muscle psoas indices measured by ultrasound in cirrhosis - Preliminary evaluation of sarcopenia assessment and prediction of liver decompensation and mortality. Dig Liver Dis. 2019 Nov;51(11):1502-1507. doi: 10.1016/j.dld.2019.08.017. Epub 2019 Sep 20. PMID 31547952
- [Background] Hida T, Ando K, Kobayashi K, Ito K, Tsushima M, Kobayakawa T, Morozumi M, Tanaka S, Machino M, Ota K, Kanbara S, Ito S, Ishiguro N, Hasegawa Y, Imagama S. <Editors' Choice> Ultrasound measurement of thigh muscle thickness for assessment of sarcopenia. Nagoya J Med Sci. 2018 Nov;80(4):519-527. doi: 10.18999/nagjms.80.4.519. PMID 30587866
- [Background] Takai Y, Katsumata Y, Kawakami Y, Kanehisa H, Fukunaga T. Ultrasound method for estimating the cross-sectional area of the psoas major muscle. Med Sci Sports Exerc. 2011 Oct;43(10):2000-4. doi: 10.1249/MSS.0b013e31821994cb. PMID 21448087
- [Background] McLean RR, Shardell MD, Alley DE, Cawthon PM, Fragala MS, Harris TB, Kenny AM, Peters KW, Ferrucci L, Guralnik JM, Kritchevsky SB, Kiel DP, Vassileva MT, Xue QL, Perera S, Studenski SA, Dam TT. Criteria for clinically relevant weakness and low lean mass and their longitudinal association with incident mobility impairment and mortality: the foundation for the National Institutes of Health (FNIH) sarcopenia project. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):576-83. doi: 10.1093/gerona/glu012. PMID 24737560
- [Background] Benz E, Trajanoska K, Lahousse L, Schoufour JD, Terzikhan N, De Roos E, de Jonge GB, Williams R, Franco OH, Brusselle G, Rivadeneira F. Sarcopenia in COPD: a systematic review and meta-analysis. Eur Respir Rev. 2019 Nov 13;28(154):190049. doi: 10.1183/16000617.0049-2019. Print 2019 Dec 31. PMID 31722892
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718